CLINICAL TRIAL: NCT05071755
Title: Gastrectomy Outcomes in Elderly Patients
Acronym: GOE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tevfik Kivilcim Uprak, Assistant Professor, Marmara University
Other Study IDs: 21s01
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Gastrectomy; Elderly; Gastric Cancer; Gastric Adenocarcinoma
Keywords: Gastrectomy; Elderly; Gastric Cancer; Prognosis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Gastrectomy — Radical Total Gastrectomy, Radical Partial gastrectomy (Proximal / Subtotal)

SUMMARY:
In this study, the investigators aimed to identify independent prognostic factors for early postoperative complications and survival in elderly patients (aged ≥65 years) with gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is the 5th most common type of cancer diagnosed worldwide and ranks 3rd in cancer-related deaths. Along with surgical resection, perioperative chemotherapy or chemoradiotherapy are the main treatment method. Various complications can be seen in the postoperative period, mainly pulmonary complications (13%), cardiac complications (6%), intra-abdominal abscesses (4%), and anastomotic leaks (3%). Approximately 5% of the patients die because of postoperative complications. It is known that low body mass index as a patient-specific factor is associated with postoperative complications and poor prognosis.

The incidence of gastric cancer remains relatively high and, with increasing life expectancy, the incidence of gastric cancer in elderly patients is increasing. Characteristics of elderly patients, such as reduced physiological function, poor nutritional status, and surgical trauma from radical gastrectomy, seem to result in higher postoperative morbidity, a longer length of hospital stays, increased healthcare costs, and higher postoperative mortality. Elderly patients may have a worse prognosis compared to younger patients, primarily because of the increased risk of postoperative complications. Perioperative nutritional support and preoperative rehabilitation are beneficial for elderly patients with gastric cancer and may reduce surgical complications and mortality. Although some studies in the literature state that radical surgery can be performed for those aged 80 and over, some studies have argued that complications increase in elderly patients and that surgery should be limited.

Aim of the study is to identify prognostic factors for postoperative outcomes in elderly patients who underwent surgery for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and older
* Operable patients with histologically confirmed gastric cancer
* Complete follow-up information

Exclusion Criteria:

* Patients under 65 years of age
* Gastric resection for non-neoplastic diseases
* Missing follow-up information

Ages: 65 Years to 100 Years | Sex: All
Age Groups: Older Adult
Study Population: The population of the research consists of patients who underwent gastrectomy with the diagnosis of gastric cancer in the General Surgery Clinic of Marmara University Pendik Training and Research Hospital, aged 65 and older between January 2014 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication rate | Within 30 days after surgery
  Complications will be reported and graded according to the Clavien-Dindo classification of surgical complications.
Postoperative mortality | Within 30 days after surgery
  Mortality during 30 days after surgery.
Overall survival | Five years
  Overall survival is defined as the time interval from the time of the radical gastrectomy to the date of all-cause death or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tevfik Uprak, MD, Principal Investigator — Marmara University Pendik Training and Research Hospital
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Araki I, Hosoda K, Yamashita K, Katada N, Sakuramoto S, Moriya H, Mieno H, Ema A, Kikuchi S, Mikami T, Watanabe M. Prognostic impact of venous invasion in stage IB node-negative gastric cancer. Gastric Cancer. 2015 Apr;18(2):297-305. doi: 10.1007/s10120-014-0362-2. Epub 2014 Apr 1. PMID 24687437
- [Background] Etoh T, Katai H, Fukagawa T, Sano T, Oda I, Gotoda T, Yoshimura K, Sasako M. Treatment of early gastric cancer in the elderly patient: results of EMR and gastrectomy at a national referral center in Japan. Gastrointest Endosc. 2005 Dec;62(6):868-71. doi: 10.1016/j.gie.2005.09.012. PMID 16301028
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Onodera T, Goseki N, Kosaki G. [Prognostic nutritional index in gastrointestinal surgery of malnourished cancer patients]. Nihon Geka Gakkai Zasshi. 1984 Sep;85(9):1001-5. Japanese. PMID 6438478